CLINICAL TRIAL: NCT02802319
Title: Ridge Preservation Following Tooth Extraction Using Porcine and Bovine Xenograft Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Brian L Mealey, Professor and Graduate Program Director, Periodontics, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC2016-0285H
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test: Porcine Xenograft (Zcore) (Experimental): Ridge preservation bone grafting surgery with porcine xenograft (Zcore)
  Interventions: Device: Porcine Xenograft (Zcore)
- Active Control: Bovine Xenograft (Bio-Oss) (Active Comparator): Ridge preservation bone grafting surgery with bovine xenograft (Bio-Oss)
  Interventions: Device: Bovine Xenograft (Bio-Oss)

INTERVENTIONS:
Device: Porcine Xenograft (Zcore) — Ridge preservation bone grafting after tooth extraction
  Arms: Test: Porcine Xenograft (Zcore)
Device: Bovine Xenograft (Bio-Oss) — Ridge preservation bone grafting after tooth extraction
  Arms: Active Control: Bovine Xenograft (Bio-Oss)

SUMMARY:
The study is a two-arm, parallel-design, randomized, prospective clinical trial designed to examine histologic wound healing following ridge preservation using bovine xenograft and porcine xenograft materials.This protocol involves procedures that are standard care. All materials are FDA-approved materials being used in an FDA-approved manner. The test group subjects will have extraction sockets grafted with porcine xenograft (Zcore). This test group will be compared to an active control group using bovine xenograft (Bio-Oss). The null hypothesis is that there will be no significant difference in formation of new vital bone between treatment groups (primary outcome).

Each subjects will have a non-molar tooth extracted and the socket grafted with either test or control graft material. At the time of dental implant placement 18-20 weeks after tooth extraction a small core biopsy specimen will be removed from the implant site. The core biopsy will then be evaluated for the primary histologic outcome of % vital bone formation and secondary histologic outcome of % residual graft material.

DETAILED DESCRIPTION:
The study is designed to examine histologic wound healing following ridge preservation using bovine xenograft and porcine xenograft materials.

This entire protocol involves procedures that are standard care. The study is a 2-arm, parallel-design, randomized, prospective clinical trial. The test group subjects will have extraction sockets grafted with porcine xenograft (Zcore). This test group will be compared to an active control group using bovine xenograft (Bio-Oss). The null hypothesis is that there will be no significant difference in formation of new vital bone between treatment groups (primary outcome).

In keeping with the protocol our study group has used several times before, the plan will be to extract non-molar teeth and graft with the test/control materials. Each subject will provide a single non-molar tooth site for study treatment. The graft material will be covered with a non-resorbable dense polytetrafluoroethylene (d-PTFE) membrane (TXT-200 singles, Osteogenics Inc). This d-PTFE membrane will be removed 4 weeks after placement during the 4-week post-op visit. Following 18-20 weeks of healing, the dental implant will be placed. To place a dental implant, an osteotomy (hole in the bone) is prepared into which the implant is placed. This osteotomy can be prepared with either a solid drill, in which case the bone that is removed is suctioned into the suction system, or with a hollow trephine drill into which a core of bone can be collected. The only "research procedure" being done in the current study is the collection of this bone core biopsy for histologic evaluation. The core biopsy will then be evaluated for the primary histologic outcome of % vital bone formation and secondary histologic outcome of % residual graft material.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included in this study if they qualify the following inclusion criteria:
* Live within 50 miles from the School of Dentistry, University of Texas Health Science Center at San Antonio
* Are able to attend a minimum of 6 visits over a 4-5 month period, as required by the study protocol
* A single rooted tooth that has been identified as requiring extraction
* Desire a dental implant to replace the missing tooth
* Have adequate restorative space for a dental implant-retained restoration
* Have at least 10mm of alveolar bone height, without impinging on the maxillary sinus or inferior alveolar canal.
* Have a dehiscence of the buccal or lingual bony plate of the tooth socket extending no more than 50% of the total depth of the socket.
* Female patients who have undergone a hysterectomy, tubal ligation, or menopause, and non-pregnant women of child-bearing potential.
* Are nonsmokers or former smokers. Current smokers may only be included if they smoke <10 cigarettes per day

Exclusion Criteria:

* Patients who live more than 50 miles from the School of Dentistry, University of Texas Health Science Center at San Antonio
* Patients who do not meet all the inclusion criteria or who will not cooperate with the required follow-up schedule.
* Patients will are mentally incompetent, prisoners, or pregnant.
* Pregnant women or women intending to become pregnant during the study period.
* Smokers who smoke >10 cigarettes per day
* Clinical and/or radiographic determinations which will preclude inclusion in this study are: Active infection other than periodontitis; Inadequate bone dimensions or restorative space for a dental implant; Presence of a disease entity, condition or therapeutic regimen which decreases probability of soft tissue and bony healing, e.g., poorly controlled diabetes, chemotherapeutic and immunosuppressive agents, autoimmune diseases, history of bisphosphonate use or long-term steroid therapy
* Positive medical history of endocarditis following oral or dental surgery.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-07; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian L Mealey, DDS, MS, Principal Investigator — UT Health Science Center at San Antonio, School of Dentistry
Locations (1):
- UT Health Science Center School of Dentistry, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lai VJ, Michalek JE, Liu Q, Mealey BL. Ridge preservation following tooth extraction using bovine xenograft compared with porcine xenograft: A randomized controlled clinical trial. J Periodontol. 2020 Mar;91(3):361-368. doi: 10.1002/JPER.19-0211. Epub 2019 Aug 23. PMID 31380563

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test: Porcine Xenograft (Zcore) | Active Control: Bovine Xenograft (Bio-Oss)
Started | 22 | 22
Completed | 20 | 17
Not Completed | 2 | 5
Not completed — Physician Decision | 2 | 1
Not completed — Lost to Follow-up | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test: Porcine Xenograft (Zcore) | Active Control: Bovine Xenograft (Bio-Oss) | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Full Range); unit: years] | 56 [24 to 79] | 58 [26 to 82] | 57 [24 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 18
  Not Hispanic or Latino | 14 | 12 | 26
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: % Vital Bone Formation (Histological)
Description: histologic determination of % vital bone formation
Time Frame: 18-20 weeks after ridge preservation
Measure: Mean (Standard Deviation); unit: % vital bone
Arm/Group | Test: Porcine Xenograft (Zcore) | Active Control: Bovine Xenograft (Bio-Oss)
Number analyzed (Participants) | 20 | 17
% vital bone | 31.27 (16.23) | 36.21 (26.51)

2. Secondary Outcome: % Residual Graft Material (Histological)
Description: histologic determination of % residual bone graft material
Time Frame: 18-20 weeks after ridge preservation
Measure: Mean (Standard Deviation); unit: % residual graft material
Arm/Group | Test: Porcine Xenograft (Zcore) | Active Control: Bovine Xenograft (Bio-Oss)
Number analyzed (Participants) | 20 | 17
% residual graft material | 19.52 (9.19) | 20.47 (15.29)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Test: Porcine Xenograft (Zcore) | Active Control: Bovine Xenograft (Bio-Oss)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/22
Other Adverse Events (participants affected / at risk) | 1/22 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test: Porcine Xenograft (Zcore) (N=22) | Active Control: Bovine Xenograft (Bio-Oss) (N=22)
Squamous cell carcinoma (Skin and subcutaneous tissue disorders) | 0 | 1 — Patient developed squamous cell carcinoma *not related to study)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test: Porcine Xenograft (Zcore) (N=22) | Active Control: Bovine Xenograft (Bio-Oss) (N=22)
fractured arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — patient had an accident and broke her arm (unrelated to study)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT02802319/Prot_SAP_000.pdf